CLINICAL TRIAL: NCT02927717
Title: An Italian Experience on Grade 3b Follicular Lymphoma
Acronym: FL3b-Oss-2015
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Barbara Botto, MD, A.O.U. Città della Salute e della Scienza
Other Study IDs: FL3b-Oss-2015
Record Dates: First submitted 2016-09-28; First posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Grade 3b Follicular Lymphoma
Keywords: Grade 3b Follicular Lymphoma; 2016 WHO Criteria; Front-line treatment; Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Study purpose is to evaluate baseline clinical data, outcome after front-line Rituximab containing chemotherapy and survival in patients with grade 3b Follicular Lymphoma.

Also an histological central review is planned in order to re-assess baseline diagnosis according to new 2016 World Health Organization (WHO) criteria.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of grade 3b Follicular Lymphoma
* Age > 18 years
* Front-line treatment with Rituximab containing chemotherapy
* Availability of histological sample for central review

Exclusion Criteria:

* Other lymphoma diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with grade 3b Follicular Lymphoma treated with Rituximab containing chemotherapy as front-line treatment
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | End of front-line treatment (evaluated from diagnosis up to 30 months)
  Number of patients who achieve Complete Response or Partial Response after treatment

SECONDARY OUTCOMES:
Progression Free Survival | From first response to last follow-up for at least 2 years (up to 15 years)
  Time from last response to nearest relapse or follow-up
Overall Survival | Date of last follow-up for at least 2 years (up to 15 years)
  Time to last follow-up or death

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Botto, MD, Principal Investigator — A.O.U. Città della Salute e della Scienza

IPD SHARING:
Plan to Share IPD: Yes
paper publication